CLINICAL TRIAL: NCT04590222
Title: Impact of a Monoamine Oxidase Inhibitor on the Phenotype of Blood Mononucleated Cells in Patients With COVID-19
Acronym: MAOi-COV19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200989; 2020-A02398-31 (Other: IDRCB)
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV2 Infection; Monoamine Oxidase Inhibitor; Activation phenotype of T and myeloid cells
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One blood sample of 60 mL (EDTA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Female, BMI≥30, mild: Females:
  Obese BMI≥30 With Mild infection n = 10
  Interventions: Other: blood sample
- Female, BMI≥30, severe: Females:
  Obese BMI≥30 With severe infection n = 10
  Interventions: Other: blood sample
- Female, BMI<30, mild: Females:
  Non-Obese BMI<30 With Mild infection n = 10
  Interventions: Other: blood sample
- Female, BMI<30, severe: Females:
  Non-Obese BMI<30 With severe infection n = 10
  Interventions: Other: blood sample
- male, BMI≥30, mild: males: Obese BMI≥30 With Mild infection n = 10
  Interventions: Other: blood sample
- male, BMI≥30, severe: males: Obese BMI≥30 With severe infection n = 10
  Interventions: Other: blood sample
- male, BMI<30, mild: males: Non-Obese BMI<30 With Mild infection n = 10
  Interventions: Other: blood sample
- male, BMI<30, severe: males: Non-Obese BMI<30 With severe infection n = 10
  Interventions: Other: blood sample
- Healthy donors from the EFS (Etablissement Français du Sang, St Louis): Healthy donors from the EFS (Etablissement Français du Sang, St Louis) including 5 men and 5 women
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — One blood sample of 60 mL (EDTA)

SUMMARY:
The principal objective is to determine the impact of phenelzine on the activation phenotype of T cells and myeloid cells during SARS-CoV2 infection

DETAILED DESCRIPTION:
Investigators want to test in vitro (in France Stage 1), and in vivo in a phase 1b/2 clinical trial (Stage 2 in Australia) a widely used antidepressant (the monoamine oxidase inhibitor (MAOi) Phenelzine (Nardil*), repurposed as an antiviral drug to treat SARS-CoV-2. Indeed this proposal leverages extensive existing data on the epigenetic mechanism of action of phenelzine and new data suggesting that it has an anti-viral action against the SARS-CoV-2 virus.

Epigenetic drugs are promising antiviral treatments capable of modifying epigenetic tags and re-programming host and viral genomes. Epigenetic modulation could be useful at least at two steps: the entry of the virus, and the regulation of the immune response. The SARS-Cov-2 depends on ACE2 and TMPRSS2 to gain cellular entry. The reduction of the expression of these proteins could therefore be protective.

Recent clinical studies have demonstrated that, in addition to their effects on neurotransmitter regulation, anti-depressants also possess anti-inflammatory characteristics via impacting pro inflammatory cytokines production which are involved in the 'cytokines storm' during severe disease. (2). These patients also have fewer circulating functional T cells and NK cells and greater numbers of dysfunctional, exhausted CD8+ T cells (3). These abnormalities are probably deleterious and reduce the efficacy of anti-viral responses.

The in-depth and patented epigenetic, cellular, and structural analyses of human cell lines harbouring the SARS-CoV-2 infective machinery and capable of propagating the virus have shown that:

* The epigenetic enzyme (histone demethylase) LSD1 directly regulates the SARS-CoV-2-binding domain of ACE2 and the protease active sites of TMPRSS2 (patented), which are critical for viral entry and propagation within the host.
* MAOi, which target LSD1 activity, inhibit the ACE2/TMPRSS2 machinery, which investigators hypothesize will prevent viral entry into the host cell to reduce viral load, disease burden, and the emergence of cytokine storms. In support of novel dual targeting viral blockage strategy recent work have shown that targeting TMPRSS2 or ACE2 alone has anti-viral activity (4).

LSD1 inhibition with Phenelzine in recent, successfully completed phase 1B clinical demonstrate that Phenelzine reverses the dysfunctional T cell phenotype and restores durable memory responses in vivo in advanced, metastatic breast cancer patients. Importantly, no adverse impact on healthy volunteer immune systems was recorded as part of the phase 1B clinical trial (5). Preclinical data shows that aged individuals have exhausted T cells compared to young individuals and MAOi re-waken these T cells resembling younger people.

Thus, investigators propose that in patients with severe COVID-19 infection, who are predominantly elderly; where dysfunctional T cells is also a feature, Phenelzine would have additional benefits on their immune function without adverse effects.

Therefore, this proposal exploits a clear mechanism of action of Phenelzine: epigenetic regulation and is the first study to explore epigenetic mechanisms in SARS-CoV-2 infection. Modulation of the epigenetism could directly counteract the virus via an antiviral effect, and indirectly via the restoration of a functional immune response.

Phenelzine has been used for nearly 60 years to treat major depressive disorder. Its side-effects, most of which are minor, are well characterized, including in the elderly or immune vulnerable.

Investigators approach is highly flexible, since LSD1 inhibition targets two immune mechanisms - a specific viral uptake pathway and the efficacy of T cell responses. Give the safety and easy applicability of Phenelzine, it lends itself to combinatorial therapeutic approaches as and when other anti-viral show efficacy. From the mechanistic perspective, investigators epigenetic approach complements and contextualises genetic studies on COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals male or female ≥18 years of age at time of enrolment
* 2.Subject (or legally authorized representative provides non opposition form prior to initiation of any study procedure.
* 3. Understands and agrees to comply with planned study procedure. (Agrees to the collection of venous blood per protocol).
* 4. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen<72hours prior to enrollment and/or a chest CT scan reported as highly likely SARS-CoV2 infection.

The different scales for severity are as follows:

* 5. Non severe patients: Clinical assessment (evidence of rales/crackles on exam) or CT scan involvement AND SpO2> 94% on room air, or ≤ 94% on room air but > 94% with nasal Oxygen with a flow rate <= 3l O2/min

For the severe infection's patients' group:

* 6. Patients requiring mechanical ventilation and/or supplemental oxygen >= 6l O2/min

For the obese patients 'group:

* 7. Obese patients will be defined as an BMI > 30
* 8. Co inclusion in non-interventional researches is possible

Exclusion Criteria:

* Pregnant and breast-feeding women
* Patients previously treated by phenelzine (Nardil®)
* Persons unable to give their no opposition
* Persons under guardianship or curatorship
* No affiliated to social insurance.
* Inclusion in interventional researches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Bicêtre Hospital (followed in hospitalization and in ambulatory services)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
levels of lymphocytes T DR + CD38 + and of monocytes CD14 dim + CD16 +. | through study completion, an average of 1 year
  evaluate the levels of the activation of T cells and myeloid cells after phenelzine exposure by the levels of the % of DR+ CD38+ T cells and CD14+dim CD16+ monocytes.

SECONDARY OUTCOMES:
level of immune checkpoints | through study completion, an average of 1 year
  evaluate the levels of the expression of immune checkpoints on T cells by flow cytometry
cytokine production and proliferation | through study completion, an average of 1 year
  evaluate the modification of functional capacities of T cells by cytokines production, and proliferation, after mitogenic and antigen recall stimulations including SARS-CoV-2 antigens
levels of neutrophils | through study completion, an average of 1 year
  assess if there is an impact of phenelzine on the activation levels of neutrophils
level of immune responses in obese patients | through study completion, an average of 1 year
  Determine if the immune responses in obese patients (a strong risk factor for severe Covid19) can be modulated in the same way compared with lean patients
level of immune responses for men and women | through study completion, an average of 1 year
  Determine if the immune responses can be modulated in the same way in men and in women (men being affected by more severe disease)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LAMBOTTE, Prof, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No